CLINICAL TRIAL: NCT03356249
Title: Next-Generation Sequencing Diagnostics of Bacteremia in Sepsis (Next GeneSiS-Trial) - Study Protocol for a Prospective, Observational, Non-interventional, Multicenter, Clinical Trial
Brief Title: Next-Generation Sequencing Diagnostics of Bacteremia in Sepsis
Acronym: NextGeneSiS
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Fraunhofer Institute for Interfacial Engineering and Biotechnology (Other); Dietmar Hopp Stiftung GmbH (Unknown)
Responsible Party: Principal Investigator, Thorsten Brenner, MD, Prof. Dr. med. Thorsten Brenner, MHBA, University Hospital, Essen
Other Study IDs: S-084/2017
Record Dates: First submitted 2017-11-19; First posted 2017-11-29 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; Next-Generation Sequencing; Bacteremia
MeSH Terms: conditions — Sepsis; Shock, Septic; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples with circulating cell-free DNA (cfDNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis Group: Patients (n=500) with suspected or proven sepsis or septic shock (according to the Sepsis-3 definitions).
  Interventions: Diagnostic Test: Next-Generation Sequencing

INTERVENTIONS:
Diagnostic Test: Next-Generation Sequencing — In 500 patients with suspected or proven sepsis or septic shock (according to the Sepsis-3 definitions), patients´ characteristics and routine blood parameters will be determined at sepsis onset as well as 72 hours afterwards. At the same time points, 2 sets of blood cultures and one blood tube for Next-Generation Sequencing (NGS)-diagnostics will be collected. An evaluation of outcome will be performed at 28 days after sepsis onset.

SUMMARY:
Sepsis remains a major challenge, even in modern intensive care medicine. The identification of the causative pathogen is crucial for an early optimization of the antimicrobial treatment regime in patients with sepsis. In this context, culture-based diagnostic procedures (e.g. blood cultures) represent the standard of care, although they are associated with relevant limitations. Therefore, culture independent methods (e.g. Next-Generation Sequencing (NGS)) seem to be an attractive alternative. By the identification of circulating cell-free DNA in the blood and the use of the quantitative sepsis indicating quantifier (SIQ) score, causing pathogens can be identified and potential contaminations can be excluded.

The goal of the presented study is therefore, to assess the diagnostic performance of a NGS-based approach for the detection of relevant infecting organisms in a big cohort of septic patients (n=500). Moreover, the plausibility of this NGS-based approach will be estimated by a panel of independent clinical specialists, retrospectively identifying potential changes in patients´ management based on NGS results.

DETAILED DESCRIPTION:
Sepsis remains a major challenge, even in modern intensive care medicine. The identification of the causative pathogen is crucial for an early optimization of the antimicrobial treatment regime in patients with sepsis. In this context, culture-based diagnostic procedures (e.g., blood cultures) represent the standard of care, although they are associated with relevant limitations. Accordingly, culture-independent molecular diagnostic procedures might be of help for the identification of the causative pathogen in infected patients. Especially the concept of an unbiased sequence analysis of circulating cell-free DNA (cfDNA) from plasma samples of septic patients by next-generation sequencing (NGS) has recently been identified to be a promising diagnostic platform for critically ill patients suffering from bloodstream infections. Although this new approach might be more sensitive and specific than culture-based state-of-the-art technologies, additional clinical trials are needed to exactly define the performance as well as clinical value of a NGS-based approach.

Next GeneSiS is a prospective, observational, non-interventional, multicenter study to assess the diagnostic performance of a NGS-based approach for the detection of relevant infecting organisms in patients with suspected or proven sepsis (according to recent sepsis definitions [sepsis-3]) by the use of the quantitative sepsis indicating quantifier (SIQ) score in comparison to standard (culture-based) microbiological testings. Moreover, the clinical value of this NGS-based approach will be estimated by a panel of independent clinical specialists, retrospectively identifying potential changes in patients´ management based on NGS results. Further subgroup analyses will focus on the clinical value especially for patients suffering from a failure of empiric treatment within the first three days after onset (as assessed by (1.) death of the patient or lack of improvement of the patient´s clinical condition (in terms of an inadequate decrease of SOFA-score) or (2.) persistent high procalcitonin levels).

This prospective, observational, non-interventional, multicenter study trial for the first time investigates the performance as well as the clinical value of a NGS based approach for the detection of bacteremia in patients with sepsis and may therefore be a pivotal step toward the clinical use of NGS in this indication.

Two sets of blood cultures (2x aerobic / 2x anaerobic) will be collected at study inclusion (=Onset) as well as 72 hours afterwards (=72h). In parallel, plasma samples for NGS-based measurements need to be obtained as described previously. Further blood samples for NGS-based measurements can be collected whenever physicians order blood cultures (2x aerobic / 2x anaerobic) because of the clinical suspicion of a bloodstream infection (BSI) within the first 3 days after study inclusion. Results of microbiological routine diagnostics in specimens different from blood (e.g. body fluid, tissue, bronchoalveolar lavage, endotracheal aspirate) will be used for further analyses when they are obtained within a timeframe of ≤72 hours prior or after the timepoints for NGS-based measurements. Clinical data collection and (if possible) PCT measurements will be performed at Onset as well as at 72h after study inclusion. The final outcome evaluation of patients will be performed at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18yr
* Informed consent
* Sepsis (with an onset ≤24h): Patients with a life-threatening organ dysfunction caused by a dysregulated host response to a suspected or proven infection. Organ dysfunction can be identified as an acute change in total SOFA score ≥2 points consequent to the infection. Patients can also be promptly identified at the bedside with qSOFA, ie, alteration in mental status, systolic blood pressure ≤100mmHg, or respiratory rate ≥22/min.
* or Septic shock (with an onset ≤24h): Patients with septic shock can be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain mean arterial pressure (MAP) ≥65mmHg and having a serum lactate level >2mmol/L (18mg/dL) despite adequate volume resuscitation.

Exclusion Criteria:

* Age ≤18yr
* Refusal to give consent
* Patient will probably be discharged from the ICU within the first 72h following inclusion
* Palliative treatment intent
* Clinician is not committed to aggressive treatment
* Death is deemed imminent and inevitable
* Patients who had previously been included, but are readmitted to the ICU during the same hospitalization, will not be included a second time.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock according to the new sepsis definitions (Sepsis-3) with an onset <24h are eligible for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity [%] (of the NGS-based SIQ-score in comparison to blood culture diagnostics, as the goldstandard for the identification of the causative pathogen in sepsis) | 2 years
  Proportion of positives that are correctly identified as such.
Specificity [%] (of the NGS-based SIQ-score in comparison to blood culture diagnostics, as the goldstandard for the identification of the causative pathogen in sepsis) | 2 years
  Proportion of negatives that are correctly identified as such.
Positive predictive value [%] (of the NGS-based SIQ-score in comparison to blood culture diagnostics, as the goldstandard for the identification of the causative pathogen in sepsis) | 2 years
  Proportion of positives that are true positive.
Negative predictive value [%] (of the NGS-based SIQ-score in comparison to blood culture diagnostics, as the goldstandard for the identification of the causative pathogen in sepsis) | 2 years
  Proportion of negatives that are true negative.
Cohen's kappa coefficient [no measuring unit; 0</=k</=1] (of the NGS-based SIQ-score in comparison to blood culture diagnostics, as the goldstandard for the identification of the causative pathogen in sepsis) | 2 years
  Measurement of the interobserver agreement between both items.

SECONDARY OUTCOMES:
Plausibility [%] (of the NGS-based SIQ-score) | 2,5 years
  Using a majority rule, SIQ-score results will be evaluated for plausibility by a panel of three independent clinical specialists not associated with the study site. Therefore, the panel will be provided with clinical case summaries, NGS results and standard-of-care results from all samples tested. Results of microbiological routine diagnostics in specimens different from blood (e.g. body fluid, tissue, bronchoalveolar lavage, endotracheal aspirate) will be included when they have been obtained within a timeframe of ≤72 hours prior or after the timepoints for NGS-based measurements.
Changes in therapy [%] (that may have occurred if the NGS-based SIQ-score had been available for clinical use) | 2,5 years
  Using a majority rule, the clinical value of the NGS-based approach will be estimated by a panel of three independent clinical specialists not associated with the study site, retrospectively identifying potential changes in patients´ management based on NGS results. Therefore, the panel will be provided with clinical case summaries, NGS results and standard-of-care results from all samples tested. Results of microbiological routine diagnostics in specimens different from blood (e.g. body fluid, tissue, bronchoalveolar lavage, endotracheal aspirate) will be included when they have been obtained within a timeframe of ≤72 hours prior or after the timepoints for NGS-based measurements. To identify potential changes in antimicrobial management that may have occurred if the results from the NGS technology had been available for clinical use, the panel will be provided with a special questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Brenner, MD, Principal Investigator — University Hospital, Essen
Locations (21):
- Germany (21):
  - RWTH Aachen University, Aachen
  - Klinikum Mittelbaden Baden-Baden Balg, Baden-Baden
  - Charité - Universitätsmedizin Berlin, Berlin
  - Evangelisches Krankenhaus Bethel gGmbH, Bielefeld
  - University Hospital Bonn, Bonn
  - Klinikum Bremerhaven Reinkenheide gGmbH, Bremerhaven
  - University Hospital Köln, Cologne
  - Duesseldorf University Hospital, Düsseldorf
  - University Hospital Essen, Essen
  - University Hospital Frankfurt, Frankfurt
  - University Medical Center Göttingen, Göttingen
  - Medical School Hannover, Hanover
  - University Hospital Heidelberg, Heidelberg
  - Kliniken Landkreis Heidenheim gGmbH, Heidenheim
  - University Hospital Leipzig, Leipzig
  - Evangelisches Krankenhaus Luckau gGmbH, Luckau
  - University Hospital rechts der Isar, Munich
  - University Hospital of Regensburg, Regensburg
  - University of Rostock, Rostock
  - University Hospital Tübingen, Tübingen
  - Ulm University Medical Center, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Decker SO, Sigl A, Grumaz C, Stevens P, Vainshtein Y, Zimmermann S, Weigand MA, Hofer S, Sohn K, Brenner T. Immune-Response Patterns and Next Generation Sequencing Diagnostics for the Detection of Mycoses in Patients with Septic Shock-Results of a Combined Clinical and Experimental Investigation. Int J Mol Sci. 2017 Aug 18;18(8):1796. doi: 10.3390/ijms18081796. PMID 28820494
- [Background] Grumaz S, Stevens P, Grumaz C, Decker SO, Weigand MA, Hofer S, Brenner T, von Haeseler A, Sohn K. Next-generation sequencing diagnostics of bacteremia in septic patients. Genome Med. 2016 Jul 1;8(1):73. doi: 10.1186/s13073-016-0326-8. PMID 27368373
- [Derived] Brenner T, Decker SO, Grumaz S, Stevens P, Bruckner T, Schmoch T, Pletz MW, Bracht H, Hofer S, Marx G, Weigand MA, Sohn K; TIFOnet Critical Care Trials Group. Next-generation sequencing diagnostics of bacteremia in sepsis (Next GeneSiS-Trial): Study protocol of a prospective, observational, noninterventional, multicenter, clinical trial. Medicine (Baltimore). 2018 Feb;97(6):e9868. doi: 10.1097/MD.0000000000009868. PMID 29419698